CLINICAL TRIAL: NCT02954601
Title: A Phase 2a, Randomized, Double-Blind, Double-Dummy, Placebo-Controlled, 3-Way Crossover Study to Compare Safety, Efficacy, and Pharmacodynamics of Single and Multiple Doses of ORMD-0801 in Adult Subjects With Type 2 Diabetes Mellitus
Brief Title: A Study of Single and Multiple Doses of Oral Insulin or Placebo in Subjects With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Oramed, Ltd. (Industry)
Collaborators: Integrium (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ORA-D-012
Record Dates: First submitted 2016-10-13; First posted 2016-11-03 (Estimated); Results first posted 2018-07-12 (Actual); Last update posted 2018-07-12 (Actual); Status verified 2018-07

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Oral Insulin; DM T2 (Diabetes Mellitus Type 2)
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — ORMD-0801; Insulin; BID protein, human; Fish Oils

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Placebo (Active Comparator): Placebo (fish oil)
  Interventions: Other: Placebo
- Dose1 (Active Comparator): Dose 1 ORMD-0801 (qd)
  Interventions: Drug: ORMD-0801 (qd)
- Dose2 (Active Comparator): Dose 2 ORMD-0801 (bid)
  Interventions: Drug: ORMD-0801 (bid)
- Dose 3 (Active Comparator): Dose 3 ORMD-0801 (tid)
  Interventions: Drug: ORMD-0801 (tid)

INTERVENTIONS:
Drug: ORMD-0801 (qd) — Dose 1 = ORMD-0801 (qd)
  Other Names: Oral Insulin
  Arms: Dose1
Drug: ORMD-0801 (bid) — Dose 2 = ORMD-0801 (bid)
  Other Names: Oral Insulin
  Arms: Dose2
Drug: ORMD-0801 (tid) — Dose 3 = ORMD-0801 (tid)
  Other Names: Oral Insulin
  Arms: Dose 3
Other: Placebo — fish oil placebo
  Other Names: fish oil
  Arms: Placebo

SUMMARY:
This is a four-way crossover (non-parallel) study with each subject receiving three of the four arms. The study will enroll approximately 30 adult subjects with T2DM from age 20 to 75 inclusive.

Following a 7-10 day Screening period, eligible subjects will enter a 3-day single-blind placebo run-in. On Day 4, each subject will be randomized to a treatment sequence that will include three treatment assignments for each of three treatment Periods according to the randomization scheme.

DETAILED DESCRIPTION:
Following the screening, eligible subjects entered a 3-day, single-blind placebo run-in. On Day 4, each subject was randomized to a treatment sequence that included three treatment assignments for each of three treatment Periods according to the randomization scheme.

Pre-assignment Details The number of participants receiving each Intervention, in each Period, is reported.

Subjects received the randomized treatment from Day 4 through Day 8. There was a 24-hour single-blind placebo washout on Day 9. Each subject received placebo for one of the three treatment periods. Each subject also received 1 of the 3 active doses randomly in each of the two other treatment periods respectively. The dosing order is random.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects, age 20 to 75 years, inclusive with type 2 diabetes mellitus.
* At Visit 2/Period 1/Day 1, subjects will have been treated for their diabetes by metformin (≥1000 mg/day; any type and regimen), metformin and a DPP-4 inhibitor ( Dipeptidyl-Peptidase)-4), metformin and an SGLT-2 (Sodium-glucose co-transporter 2) inhibitor, metformin and TZD (Thiazolidinediones), or metformin and sulfonylurea. Subjects will have been on a stable regimen of metformin (defined as the same metformin dose and type) and other treatments for at least 8 weeks prior to Visit 2/Period 1/Day 1.
* Body Mass Index (BMI) between 25 and 40 kg/m2, inclusive, at Screening.
* Hemoglobin A1c (HbA1c) between ≥7.5 and ≤10.5% at Screening.
* Fasting serum glucose greater than or equal to 126 mg/dL at Screening.
* Females of childbearing potential must have a negative serum pregnancy test result at Screening and a negative urine pregnancy test at Visit 2/Day 1 for all study Periods.
* Females who are not of childbearing potential are defined as:

  i. Postmenopausal (defined as at least 12 months with no menses in women ≥45 years of age) ii. Has had a hysterectomy and/or bilateral oophorectomy, bilateral salpingectomy, or bilateral tubal ligation/occlusion at least 6 weeks prior to screening; OR iii. Has a congenital or acquired condition that prevents childbearing.
* Females of childbearing potential agree to avoid becoming pregnant while receiving study treatment and for 14 days after the last dose of study treatment by complying with one of the following:

  i. practice abstinence† from heterosexual activity OR ii. Use (or have her partner use) acceptable contraception during heterosexual activity.

Exclusion Criteria:

* Usage of anti-diabetic agents other than metformin, sulfonylurea, SGLT-2 inhibitors, TZD, or DPP-4 inhibitors within 6 weeks prior to Visit 2/Period 1/Day 1.
* Presence of any clinically significant endocrine disease according to the Investigator (euthyroid subjects on replacement therapy will be included if the dosage of thyroxine is stable for at least six weeks prior to Screening).
* Clinical diagnosis of type 1 diabetes.
* Fasting serum glucose >300 mg/dL at Screening; a single repeat test is allowable.
* Evidence of unawareness of hypoglycemia, a documented plasma glucose ≤50 mg/dL in the absence of symptoms of hypoglycemia at Screening.
* Presence of any clinically significant condition (in the opinion of the Investigator) that might interfere with the evaluation of study medication, such as significant renal, hepatic, gastrointestinal (GI), cardiovascular (CV), immune disease, blood dyscrasias or any disorders causing hemolysis or unstable red blood cells, or clinically important hematological disorders (i.e. aplastic anemia, myeloproliferative or myelodysplastic syndromes, thrombocytopenia) at Screening.
* Presence or history of cancer within the past 5 years of Screening, with the exception of adequately-treated localized basal cell skin cancer or in situ uterine cervical cancer.

  1. A subject with a history of malignancy >5 years prior to Screening should have no evidence of residual or recurrent disease.
  2. A subject with a history of melanoma, leukemia, lymphoma, or renal carcinoma is excluded.
* Laboratory abnormalities at Screening including:

  1. C-peptide < 1.0 ng/mL;
  2. Positive pregnancy test in females of childbearing potential (at Screening and Visit 2/Periods 1-3/Day 1);
  3. Abnormal serum thyrotropin (TSH) levels below the lower limit of normal or >1.5X (1.5 times) the upper limit of normal
  4. Elevated liver enzymes (alanine transaminase (ALT), alanine aminotransferase (AST), alkaline phosphatase) >2X the upper limit of normal.
  5. Very high triglyceride levels (>600 mg/dL); a single repeat test is allowable.
  6. Any relevant abnormality that would interfere with the efficacy or the safety assessments during study treatment administration.
* Positive history of active liver disease (other than non-alcoholic hepatic steatosis), including chronic hepatitis B or C, primary biliary cirrhosis, or active symptomatic gallbladder disease.
* Positive history of HIV.
* Use of the following medications:

  1. History of use of insulin for more than 1 week within 6 months prior to and none within 6 weeks prior to Visit 2/Period 1/Day 1.
  2. History of use of aprotinin at any time prior to Screening (e.g., Trasylol, any type or dose).
  3. Administration of thyroid preparations or thyroxine (except in subjects on stable replacement therapy) within 6 weeks prior to Screening.
  4. Administration of systemic long-acting corticosteroids within two months or prolonged use (more than one week) of other systemic corticosteroids or inhaled corticosteroids (if daily dosage is > 1,000 μg equivalent beclomethasone) within 30 days prior to Screening. Intra-articular and/or topical corticosteroids are not considered systemic.
  5. Use of medications known to modify glucose metabolism or to decrease the ability to recover from hypoglycemia such as oral, parenteral, and inhaled steroids (as discussed above), and immunosuppressive or immunomodulating agents.
* Subject is on a weight loss program and is not in the maintenance phase, or subject has started weight loss medication (e.g., orlistat or liraglutide), within 8 weeks prior to Screening. Subjects who have had bariatric surgery are also excluded.
* Subject is pregnant or breast-feeding.
* Subject has a Screening systolic blood pressure ≥165 mmHg or diastolic blood pressure ≥100 mmHg. Subjects will be allowed to take a BP rescue medication.
* Subject is a user of recreational or illicit drugs or has had a recent history (within 1 year of Screening) of drug or alcohol abuse or dependence. (Note: Alcohol abuse includes heavy alcohol intake as defined by >3 drinks per day or >14 drinks per week, or binge drinking) at Screening.
* Any clinically significant ECG abnormality at Screening or cardiovascular disease. Clinically significant cardiovascular disease will include:

  1. History of stroke, transient ischemic attack, or myocardial infarction within 6 months prior to Screening,
  2. History of or currently have New York Heart Associate Class II-IV heart failure prior to Screening, or
* One or more contraindications to metformin.
* At the Principal Investigator's discretion, any condition or other factor that is deemed unsuitable for subject enrollment into the study.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2016-10; Primary Completion 2017-02-24 (Actual); Study Completion 2017-03-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joel M Neutel, M. D., Principal Investigator — Orange County Research Center
Locations (1):
- Orange County Research Center, Tustin, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Following the screening, eligible subjects entered a 3-day, single-blind placebo run-in. On Day 4, each subject was randomized to a treatment sequence for each of three treatment periods, each period was either placebo or 1 of the 3 treatments). All subjects received placebo and only 2 of the 3 treatments.
Pre-assignment Details: The number of participants receiving each intervention, in each Period, is reported. In each treatment period, each subject received randomly either placebo, qd, bid, or tid for each of 3 treatment periods. Subjects received the randomized treatment from Day 4 through Day 8. There was a 24-hour single-blind placebo washout on Day 9.
Groups:
- Placebo: Placebo (fish oil) Placebo: fish oil placebo
- Dose1: Dose 1 = ORMD-0801 qid
- Dose2: Dose 2 = ORMD-0801 bid
- Dose 3: Dose 3 = ORMD-0801 tid
Period: First Intervention (Five Days)
Arm/Group | Placebo | Dose1 | Dose2 | Dose 3
Started | 11 | 6 | 8 | 7
Completed | 11 | 6 | 7 | 7
Not Completed | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0
Period: Second Intervention (Five Days)
Arm/Group | Placebo | Dose1 | Dose2 | Dose 3
Started | 11 | 6 | 8 | 6
Completed | 11 | 6 | 8 | 6
Not Completed | 0 | 0 | 0 | 0
Period: Third Intervention (Five Days)
Arm/Group | Placebo | Dose1 | Dose2 | Dose 3
Started | 9 | 8 | 6 | 8
Completed | 9 | 8 | 6 | 8
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: ITT Population
Groups:
- ORMD-0801 qd: Oral Insulin once per day
- ORMD-0801 Bid: Oral Insulin twice per day
- ORMD-0801 Tid: Oral Insulin three times per day
- Total: Total of all reporting groups
Arm/Group | Placebo | ORMD-0801 qd | ORMD-0801 Bid | ORMD-0801 Tid | Total
Number analyzed (Participants) | 11 | 6 | 7 | 7 | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.27 (7.00) | 57.17 (11.37) | 59.5 (7.03) | 58.71 (7.54) | 57.72 (7.77)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 5 | 1 | 3 | 12
  Male | 8 | 1 | 6 | 4 | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 3 | 4 | 6 | 17
  Not Hispanic or Latino | 7 | 3 | 3 | 1 | 14
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 1 | 1 | 0 | 4
  White | 9 | 5 | 5 | 6 | 25
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Child-Bearing Status [Count of Participants; unit: Participants]
  Not Applicable (Male) | 8 | 1 | 6 | 4 | 19
  Of Childbearing Potential | 0 | 0 | 0 | 0 | 0
  Post Hysterectomy | 1 | 1 | 0 | 2 | 4
  Surgically Sterilized | 0 | 2 | 0 | 0 | 2
  At least 1 year Post-Menopausal | 2 | 2 | 1 | 1 | 6
Alcohol History [Count of Participants; unit: Participants]
  Never | 6 | 3 | 2 | 5 | 16
  Current | 5 | 3 | 4 | 2 | 14
  Former | 0 | 0 | 1 | 0 | 1
Tobacco History [Count of Participants; unit: Participants]
  Never | 8 | 5 | 5 | 5 | 23
  Current | 1 | 0 | 0 | 1 | 2
  Former | 2 | 1 | 2 | 1 | 6
Caffiene History [Count of Participants; unit: Participants]
  Never | 1 | 1 | 1 | 1 | 4
  Current | 10 | 5 | 6 | 5 | 26
  Former | 0 | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change in Glucose Levels Between Pre-treatment and End of Treatment as Measured by 24-hour Continuous Glucose Monitoring (CGM)
Description: Measure the change in Glucose (mg/dL) by 24 hour CGM between Day3 and Day8 (Change in mg/dL between run-in and Day 5 of Active treatment)
Time Frame: Day 3 (run-in) and Day 8 (Day 5 of Active treatment)
Population: Intend to Treat Population
Measure: Mean (Standard Deviation); unit: mg/dL
Groups:
- Dose 1: ORMD-0801 qid
- Dose 2: ORMD-0801 bid
- Dose 3: ORMD-0801 tid
Arm/Group | Placebo | Dose 1 | Dose 2 | Dose 3
Number analyzed (Participants) | 31 | 20 | 20 | 21
mg/dL | -4.94 (4.418) | -10.00 (7.236) | -1.21 (7.397) | -11.42 (8.451)
Statistical Analysis 1: Comparison: Placebo vs Dose 1 vs Dose 2 vs Dose 3; Test type: Other — Values obtained using a Mixed Model Repeated Measures Analysis of Variance with an unstructured covariance matrix. Treatment, Period and Baseline value (for change and percent change) are factors in the model with repeated values for a subject; p = 0.1311, Mixed Models Analysis

2. Secondary Outcome: Calculate the C-peptide Ratio for Single and Multiple Doses of ORMD-0801 vs Placebo.
Description: For each dose, calculate the ratio of the C-Peptide measurement area-under-the-curve (ng-hr/mL) Day 8 to the C-peptide measurement area-under-the-curve (ng-hr/mL) Day 3. This ratio is called the C-peptide Ratio.
Time Frame: Day 3 and Day 8
Population: Intend to Treat (ITT)
Measure: Mean (Standard Error); unit: ratio
Arm/Group | Placebo | Dose 1 | Dose 2 | Dose 3
Number analyzed (Participants) | 31 | 20 | 21 | 21
ratio | 0.97 (0.034) | 1.01 (0.056) | 1.03 (0.047) | 0.93 (0.051)

3. Secondary Outcome: The Number Hypoglycemic Events for Single and Multiple Doses of ORMD-0801 vs Placebo
Description: The number of safety parameter hypoglycemic events for single and multiple doses of ORMD-0801 vs placebo.
Time Frame: Day 3 through Day 8 of treatment
Population: Safety population
Measure: Number; unit: number of hypoglycemic events
Arm/Group | Placebo | Dose 1 | Dose 2 | Dose 3
Number analyzed (Participants) | 31 | 20 | 21 | 21
number of hypoglycemic events | 3 | 2 | 4 | 5

4. Secondary Outcome: Calculate the Difference Between Values of Pre-treatment and End-of-treatment Mean Daytime CGM Glucose
Description: Calculate the difference between pre-treatment (Day 3) and end of treatment (Day 8) mean daytime CGM glucose for single and multiple doses of ORMD-0801 vs placebo.
Time Frame: Day 3 and Day 8 (two timepoints)
Population: Intend to Treat mean values reported for Doses 1, 2, and 3 are placebo-adjusted doses (Active dose mean minus placebo dose mean)
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo | Dose 1 | Dose 2 | Dose 3
Number analyzed (Participants) | 31 | 20 | 21 | 20
mg/dL | -4.11 (5.080) | -13.96 (7.775) | 1.13 (7.772) | -16.78 (8.613)
Statistical Analysis 1: Comparison: Placebo vs Dose 1 vs Dose 2 vs Dose 3; Values obtained using a Mixed Model Repeated Measures Analysis of Variance with an unstructured covariance matrix. Treatment period and Baseline value (for change and percent change) are factors in the model with repeated values for subject; Test type: Other; p = 0.3061, Mixed Models Analysis

ADVERSE EVENTS:
Time Frame: One Year
Groups:
- Dose 1: Dose 1 = ORMD-0801 qid
- Dose 2: Dose 2 = ORMD-0801 bid
Arm/Group | Placebo | Dose 1 | Dose 2 | Dose 3
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/20 | 0/21 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/20 | 0/21 | 0/20
Other Adverse Events (participants affected / at risk) | 12/31 | 7/20 | 11/21 | 3/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=31) | Dose 1 (N=20) | Dose 2 (N=21) | Dose 3 (N=20)
Hypoglycemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 4 (4) | 1 (1) — Number of Hypoglycemic events during treatment period
Gastrointestinal disorders (Gastrointestinal disorders) | 3 (3) | 1 (1) | 2 (2) | 0 (0)
Eye Disorders (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Metabolism and Nutrional Disorders (Metabolism and nutrition disorders) | 7 (7) | 5 (5) | 6 (6) | 2 (2)
Muskuloskeletal and connective tissue disorders (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Nervous System Disorders (Nervous system disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2016-08-23): https://cdn.clinicaltrials.gov/large-docs/01/NCT02954601/Prot_000.pdf
  • Statistical Analysis Plan (2017-01-05): https://cdn.clinicaltrials.gov/large-docs/01/NCT02954601/SAP_001.pdf